CLINICAL TRIAL: NCT02510287
Title: A Comparison of Epidural Analgesia: Continuous Infusion Versus Programmed Intermittent Boluses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Santa Fe de Bogota (Other)
Responsible Party: Principal Investigator, Leopoldo Ferrer, MD anesthesiologist, Fundación Santa Fe de Bogota
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CCEI-3413-2015
Record Dates: First submitted 2015-07-22; First posted 2015-07-29 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Labor Pain
Keywords: analgesia, epidural; labor pain; patient satisfaction
MeSH Terms: conditions — Labor Pain; Agnosia; Patient Satisfaction | interventions — Bupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Continuous Epidural Infusion (Active Comparator): 1. An initial dose of 10 ml of 0.1% bupivacaine (2 ml of 0.5% bupivacaine and 50 mcg / ml fentanyl in 7 ml of normal saline solution) will be given.
  2. A continuous infusion of 0.1% bupivacaine and fentanyl 2 mcg / ml (8-12 ml / hour) will then be administered.
  3. Upon patient request, rescue bolus of 8-10 ml of 0.1% bupivacaine will be administered.
  4. If needed, during the second phase (9-10 centimeters of cervical dilation) a 2% lidocaine without epinephrine (8-10 cc) bolus will be administered.
  Interventions: Drug: Bupivacaine and Fentanyl Initial Dose; Drug: Bupivacaine and Fentanyl: Continuous Epidural Infusion; Drug: Rescue Bolus; Drug: Lidocaine
- Programmed Intermittent Epidural Bolus (Experimental): 1. An initial dose of 10 ml of 0.1% bupivacaine (2 ml of 0.5% bupivacaine and 50 mcg / ml fentanyl in 7 ml of normal saline solution) will be given.
  2. A 0.1% bupivacaine and fentanyl 2 mcg / ml (8-12ml) bolus will be administered each hour at a rate of 500ml/hour.
  3. Upon patient request, rescue bolus of 8-10 ml of 0.1% bupivacaine will be administered.
  4. If needed, during the second phase (9-10 centimeters of cervical dilation) a 2% lidocaine without epinephrine (8-10 cc) bolus will be administered .
  Interventions: Drug: Bupivacaine and Fentanyl Initial Dose; Drug: Bupivacaine and Fentanyl: Programmed Intermittent Epidural Bolus; Drug: Rescue Bolus; Drug: Lidocaine

INTERVENTIONS:
Drug: Bupivacaine and Fentanyl Initial Dose — 10 ml of 0.1% bupivacaine (2 ml of 0.5% bupivacaine and 50 mcg / ml fentanyl in 7 ml of normal saline solution)
Drug: Bupivacaine and Fentanyl: Continuous Epidural Infusion — 0.1% bupivacaine and fentanyl 2 mcg / ml (8-12 ml / hour)
  Arms: Continuous Epidural Infusion
Drug: Bupivacaine and Fentanyl: Programmed Intermittent Epidural Bolus — A 0.1% bupivacaine and fentanyl 2 mcg / ml (8-12ml) bolus will be administered each hour at a rate of 500ml/hour
  Arms: Programmed Intermittent Epidural Bolus
Drug: Rescue Bolus — Upon patient request, rescue bolus of 8-10 ml of 0.1% bupivacaine will be administered.
Drug: Lidocaine — If needed, during the second phase (9-10 centimeters of cervical dilation) a 2% lidocaine without epinephrine (8-10 cc) bolus will be administered.

SUMMARY:
The analgesic approach in labor can be done in different ways, among which the neuraxial approach has shown the best analgesic results and fetal outcomes. Currently, programmed epidural intermittent bolus has been included in the neuraxial approach for a better distribution of the solution into the epidural space as compared with the continuous infusion strategy. In this study, the investigators seek to compare both strategies in 132 laboring women.

ELIGIBILITY:
Inclusion Criteria:

* At term pregnancy
* Laboring patients requiring epidural analgesia

Exclusion Criteria:

* American Society of Anesthesiologists physical status > or equal than 3
* allergy to local anesthesics
* Neuraxial contraindications
* Hemodynamic instability
* Systemic disease such as diabetes mellitus or hypertension
* Chronic usage of analgesics
* Disease associated to pregnancy such as gestational diabetes, preeclampsia, fetal malformations among others

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2015-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pain level in laboring women measured by the Numeric Analog Scale | one year
  to compare pain level in each arm once epidural analgesia is applied until birth

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Santa Fe, Bogotá, Bogota D.C., Colombia